CLINICAL TRIAL: NCT00268138
Title: Phase 4 Study Prevention of Incipient Carious Lesions (White Spot Lesions) in Patients With Fixed Orthodontic Appliances Following the Application of Elmex Gel
Brief Title: Elmex Gel Efficacy in Preventing White Spot Lesions
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Gaba International AG (Industry)
Responsible Party: Dr Meir Redlich, Hadassah
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 123456-HMO-CTIL
Record Dates: First submitted 2005-12-21; First posted 2005-12-22 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2005-12

CONDITIONS: Dental Caries
Keywords: amine fluoride; white spot lesions; qlf
MeSH Terms: conditions — Dental Caries | interventions — Fluorides

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: elmex gel — elmex gel once a week
  Other Names: fluoride

SUMMARY:
the objective of this phase IV study: to establish the efficacy of elmex gel with a fluoride concentration of 1.25% compared with placebo by determining prevention of white spot lesions in patients wearing fixed orthodontic appliances.

DETAILED DESCRIPTION:
314 healthy subjects undergoing orthodontic treatment will be examined. follow up will take place from bonding the appliance till debonding, at least 12 months and no more than 30 months.

tooth brushing with product (test product or control) once per week during the entire study.

4 times a year additional tray application of test product or control. subjects wiil clean their teeth with the toothpaste they usually use during the entire study.

toothbrush and a sandglass will be provided every 6 weeks

ELIGIBILITY:
Inclusion Criteria:

* treatment plan: minimum of 10 teeth to be bonded labially at least 10 years old
* written declaration of informed consent

Exclusion Criteria:

* known allergy to components of test products
* handicapped patients who have difficulties brushing their teeth
* pathological desquamation changes
* known pregnancy, breast feeding
* eating disorders
* disease that effect dental hard tissue
* participation in another clinical trial either currently or within the lase 30 days

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 314 (Estimated)
Dates: Start 2006-04; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
time and frequency of visually detected WSL (white spot lesions) | 3 month

SECONDARY OUTCOMES:
mineral loss according to QLF readings | 3 month
Frequency and chronoloy of WSL | 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Meir Redlich, DMD PhD, Principal Investigator — Hadassah Medical Center, Dept of Orthodontics; Paul George Jost-Brinkmann, Prof, Principal Investigator — Charite - Berlin, Dept of Orthodontics, Center of Dentistry
Locations (2):
- Charite University, Berlin, Germany
- Hadassah Medical Organization, Jerusalem, Israel, Jerusalem, Israel